CLINICAL TRIAL: NCT01239914
Title: CathOlic Medical Center percutAneous Coronary inTervention Registry (COACT)
Acronym: COACT
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Collaborators: Seoul St. Mary's Hospital (Other); Yeouido St. Mary's Hospital (Other); Bucheon St. Mary's Hospital (Other); St.Paul's Hospital, Korea (Other); Incheon St.Mary's Hospital (Other); Saint Vincent's Hospital, Korea (Other); Daejeon St. Mary's hospital (Other)
Responsible Party: Principal Investigator, Kiyuk Chang, MD,PhD, Professor, The Catholic University of Korea
Other Study IDs: COACT
Record Dates: First submitted 2010-11-12; First posted 2010-11-15 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Drug Eluting Stent; Coronary Artery Disease; Polymorphism; Cholesterol; Biomarker
Keywords: drug eluting stent; coronary artery disease; Korean registry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood, serum and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
COACT registry is a multicenter registry of consecutive patients undergoing coronary stent implantation at 8 centers in the Catholic University of Korea to evaluate the real world management of patients with coronary artery disease and to assess their in-hospital, medium and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients who underwent percutaneous coronary intervention
* written informed consent for the DNA and serum databank

Exclusion Criteria:

* patients who did not agreed to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all comers who admitted cardiovascular center for coronary stent implantation
Sampling Method: Non-Probability Sample
Enrollment: 11719 (Actual)
Dates: Start 2005-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
All causes mortality | 6month, each year
Cardiac death | 6 month, each year
Myocardial infarction | 6 month, each year
target lesion revascularization | 6 month, each year
target vessel revascularization | 6 month, each year

SECONDARY OUTCOMES:
non target vessel revascularization | 6 month, each year
Stent thrombosis | 6 month, each year
Serum databank for evaluation of biomarkers outcomes | 6 month, each year
Pharmacogenetic and cardiovascular genetic studies associated to clinical outcomes | 6 month, each year

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bae Seung, M.D.,PhD, Study Chair — Seoul St. Mary's Hospital
Locations (8):
- South Korea (8):
  - Bucheon St.Mary Hospital, Bucheon-si, Gyeonggido
  - St.Vincent's Hospital, Suwon, Gyeonggido
  - Uijeongbu St.Mary's Hospital, Uijeongbu-si, Gyeonggido
  - Daejeon St.Mary's Hospital, Daejeon
  - Incheon St.Mary's Hospital, Incheon
  - Seoul St.Mary's Hospital, Seoul
  - St.Paul's Hospital, Seoul
  - Yeouido St.Mary Hospital, Seoul

REFERENCES:
- [Derived] Kim HS, Chang K, Koh YS, Park MW, Choi YS, Park CS, Oh M, Kim EY, Shon JH, Shin JG, Seung KB. CYP2C19 poor metabolizer is associated with clinical outcome of clopidogrel therapy in acute myocardial infarction but not stable angina. Circ Cardiovasc Genet. 2013 Oct;6(5):514-21. doi: 10.1161/CIRCGENETICS.113.000109. Epub 2013 Sep 9. PMID 24019397